CLINICAL TRIAL: NCT05278338
Title: A Multicenter, Randomized, Double-blind, Placebo/Positive-controlled Phase II Study to Evaluate the Efficacy and Safety of JMT103 in Postmenopausal Women With Osteoporosis
Brief Title: Efficacy and Safety of JMT103 in the Treatment of Postmenopausal Women With Osteoporosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMT103-CSP-008
Record Dates: First submitted 2022-03-08; First posted 2022-03-14 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group a (Experimental): JMT103 45 mg
  Interventions: Drug: JMT103
- Group b (Experimental): JMT103 60 mg
  Interventions: Drug: JMT103
- Group c (Experimental): JMT103 90 mg
  Interventions: Drug: JMT103
- Group d (Active Comparator): Denosumab 60 mg
  Interventions: Drug: Denosumab
- Group e (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMT103 — subcutaneous injection, once every 6 months (Q6M), with a total of 2 administrations
  Arms: Group a; Group b; Group c
Drug: Denosumab — subcutaneous injection, once every 6 months (Q6M), with a total of 2 administrations
  Arms: Group d
Drug: Placebo — subcutaneous injection, once every 6 months (Q6M), with a total of 2 administrations
  Arms: Group e

SUMMARY:
This study is to evaluate the efficacy and safety of JMT103 in the treatment of postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo/positive-controlled Phase II clinical study to evaluate the efficacy, safety, immunogenicity and pharmacokinetic characteristics of JMT103 in the treatment of postmenopausal women with osteoporosis. Subjects will be screened within -28 days before treatment, and subjects who meet the inclusion/exclusion criteria will be included in the study. The enrolled postmenopausal women with osteoporosis who meet the diagnostic criteria for osteoporosis will be randomized in a 1:1:1:1:1 ratio into Test Group a (JMT103 45 mg group), Test Group b (JMT103 60 mg group), Test Group c (JMT103 90 mg group), Control Group d (denosumab 60 mg group) and Control Group e (placebo group). JMT103,denosumab and placebo will be administered as a single subcutaneous (SC) injection at the beginning of the treatment phase and at 6 months following the initial dose. Each subject will be followed up for 12 months after the first administration. Throughout the research process, subjects will be required to supplement ≥1000 mg of calcium and ≥800 IU of vitamin D every day.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, capable of autonomous action, aged 50-85 years (inclusive);
2. Menopause is defined as menopause for ≥2 years, which can be spontaneous amenorrhea for ≥2 years or bilateral oophorectomy for ≥2 years. If bilateral oophorectomy status is unknown, the follicle stimulating hormone (FSH) level should be greater than or equal to 40 mIU/mL to confirm the menopausal status;
3. Meet the diagnostic criteria for osteoporosis: Based on the results of BMD measurement by dual-energy X-ray absorptiometry (DXA), lumbar spine (mean BMD of L1-L4 or more than 2 measurable vertebral bodies), total hip or femur neck BMD is -4.0 ≤ T-value ≤ -2.5; or lumbar spine, total hip or femoral neck BMD is -2.5 < T-value < -1.0 and a history of fragility fractures of the proximal humerus, pelvis or distal forearm; or a history of fragility fractures of the hip or vertebral bodies;
4. The subject can maintain good communication with the investigator and comply with the various requirements of the clinical trial, and is expected to be able to complete the entire trial process;
5. Be able to be fully informed and sign an informed consent form.

Exclusion Criteria:

1. A history of fractures of more than 2 vertebral bodies;
2. Subjects with bone metabolic diseases other than osteoporosis: a. various metabolic bone diseases, such as osteomalacia or osteogenesis imperfecta, as these diseases may interfere with the study results; b. Paget's disease; c. Cushing syndrome; d. hyperprolactinemia; e. others;
3. Currently suffering from hyperparathyroidism or hypoparathyroidism;
4. Hyperthyroidism or hypothyroidism. Subjects with hypothyroidism on stable (for at least 3 months) thyroid hormone replacement therapy can be selected, but the following conditions must be met: a. If the TSH level is below the normal range, the subject cannot participate in the study. b. If the TSH level is elevated (>5.5 μIU/mL but ≤10.0 μIU/mL), serum T4 should be measured. If the serum T4 is in the normal range, the subject can be selected. If the serum T4 is outside the normal range, the subject cannot participate in the study. c. If the TSH level is greater than 10.0 μIU/mL, the subject cannot participate in the study;
5. Rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus and other rheumatic immune diseases;
6. Malabsorption syndrome: Malabsorption syndrome or various gastrointestinal diseases related to malabsorption, such as Crohn's disease and chronic pancreatitis;
7. Previously or currently suffering from osteomyelitis or osteonecrosis of the jaw; dental surgery or oral surgery wounds that have not healed; acute dental or jaw disease requiring oral surgery; those who have planned to undergo invasive dental surgery during the study period;
8. Liver disease: a. liver cirrhosis; b. unstable liver disease (defined as ascites, hepatic encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice); c. known or clinically significant biliary tract abnormalities judged by the investigator (except Gilbert syndrome, asymptomatic gallstones and gallbladder polyps);
9. Uncontrolled concomitant diseases, including but not limited to: uncontrolled diabetes (>grade 2, NCI-CTCAE 5.0), symptomatic congestive heart failure, hypertension (blood pressure is still ≥150/90 mmHg after standard treatment), unstable angina, sick sinus syndrome (>grade 2, NCI-CTCAE 5.0), severe arrhythmia, history of myocardial infarction within the past 6 months and echocardiogram showing left ventricular ejection fraction <50%;
10. Active bacterial or fungal infection requiring systemic treatment within 7 days before randomization;
11. Those with active hepatitis B [HBsAg positive with HBV-DNA exceeding 1000 copies/mL (500 IU/mL) or higher than the lower limit of detection, whichever is lower]; subjects with active hepatitis C (HCV antibody positive with HCV-RNA level higher than the upper limit of detection); HIV antibody or syphilis antibody positive;
12. Those who are known to have active tuberculosis (TB) or suspected of active TB;
13. Those with malignant tumors within 5 years before screening, except for tumors that are expected to be cured after treatment (such as completely resected basal cell carcinoma or squamous cell carcinoma, cervical cancer or ductal carcinoma of the breast in situ, etc.);
14. Those who have used intravenous bisphosphonates, fluorides or strontium agents for the treatment of osteoporosis in the last 5 years (from the signing of the informed consent form), or oral bisphosphonates for the treatment of osteoporosis (from the date of signing the informed consent form): a. those with cumulative use greater than or equal to 3 years cannot be selected; b. those with cumulative use greater than 3 months but less than 3 years, and the last dose administered within 1 year before the date of signing the informed consent form cannot be selected (those whose last dose was one year or more before the date of signing the informed consent form can be selected); c. those with cumulative use less than or equal to 3 months can be selected;
15. Those who have used anti-receptor activator of nuclear factor-κB ligand (RANKL) antibody within one year before prior screening;
16. Those who have received drugs that affect bone metabolism within 3 months before screening: a. parathyroid hormone (PTH) or PTH derivatives, such as teriparatide; b. anabolic hormones or testosterone; c. glucocorticoids (equivalent to daily use > 5 mg of prednisone > 10 days); d. sex hormone replacement therapy; e. selective estrogen receptor modulators (SERM), such as raloxifene; f. calcitonin, calcitriol or vitamin D derivatives (cumulative use> 30 days, and used within 6 weeks before the signing of the informed consent form); g. other bone active drugs including anticonvulsants (except benzodiazepines) and heparin; h. long-term systemic use of ketoconazole, adrenocorticotropic hormone (ACTH), cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, or gonadotropin releasing hormone agonists;
17. Currently receiving other clinical study drugs, and the last dose administered less than 4 weeks or 5 elimination half-lives (t1/2) from the date of study drug administration (whichever is longer);
18. Those known to have allergies or hypersensitivity to JMT103 formulations, control drugs, calcium and vitamin D preparations;
19. Those who have received the COVID-19 vaccine within 4 weeks before administration;
20. Those whose blood system, liver and kidney function, and coagulation system examinations meet the following conditions:

    * Blood system (without receiving blood transfusion or hematopoietic stimulating factor treatment within 7 days before the signing of the informed consent form): absolute neutrophil value (ANC) <1.5×10^9/L; platelet (PLT) <75×10^9/L; hemoglobin (Hb) <90 g/L;
    * Liver function: total bilirubin (TBIL)>1.5×upper limit of normal (ULN), alanine aminotransferase (ALT)>2.5×ULN (subjects are allowed to be retested after a rest for 2-4 weeks; if the retest shows ALT<2.5×ULN, they can be included in this study), aspartate aminotransferase (AST)> 2.5×ULN; for subjects with liver metastasis or liver cancer: TBIL>3×ULN, ALT>5×ULN, and AST> 5×ULN;
    * Kidney function: urine protein ≥2+ or 24-hour urine protein quantitation ≥1.0 g; creatinine clearance* (CrCl) calculated value <60 mL/min;
    * Coagulation function: activated partial thromboplastin time: (APTT)>1.5×ULN; international normalized ratio (INR)>1.5×ULN;
21. Vitamin D deficiency: 25-(OH) vitamin D <20 ng/mL. Subjects are allowed to receive vitamin D 5000 IU/day for supplementation, and take a retest after 4-6 weeks. If 25-(OH) vitamin D is retested to be >20 ng/mL, the subjects can be enrolled;
22. Blood calcium abnormalities: current hypocalcemia or hypercalcemia. Serum calcium or serum calcium corrected for albumin is ≤2.2 mmol/L (8.8 mg/dL) or ≥2.9 mmol/L (11.5 mg/dL); subjects are not allowed to use calcium supplements at least 8 hours before blood draw for serum calcium screening determination; Conditions that affect the determination of bone mineral density by dual-energy
23. Conditions that affect the determination of BMD by dual-energy X-ray absorptiometry: less than 2 measurable lumbar vertebral bodies; height, weight, or waist circumference that may hinder accurate measurement; severe scoliosis and other conditions that affect BMD testing;
24. Subjects who are judged by the investigator to be at high risk of fractures and must receive active drug treatment;
25. Subjects who are judged by the investigator to be unsuitable for inclusion in the study.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change rate of lumbar bone mineral density (BMD) from baseline at 12 months of JMT103 treatment | Baseline and 12 months
  Dual-energy X-ray absorptiometry (DXA) will be performed to measure the bone mineral density of the subject's lumbar spine (the mean BMD of L1-L4 or more than 2 measurable vertebral bodies), the total hip and the femoral neck during the screening period, and at 3 months, 6 months and 12 months after the first administration and early withdrawal. Bone mineral density will be assessed centrally by DXA.

SECONDARY OUTCOMES:
Change rate of lumbar spine BMD from baseline at 6 months of JMT103 treatment | Baseline and 6 months
Change rate of total hip and femoral neck BMD from baseline at 12 months of JMT103 treatment | Baseline and 12 months
Change rate of serum type I collagen cross-linked C-terminal peptide (s-CTX) from baseline at 1, 3, 6 and 12 months of treatment | Day 1,15,29 and 3,6,12 months
  In this study, the central laboratory will be entrusted with the testing of biomarker samples. About 3.5 mL of venous whole blood will be collected each time.
Change rate of type I procollagen N-terminal propeptide (PINP) from baseline at 1, 3, 6 and 12 months of treatment | Day 1,15,29 and 3,6,12 months
  In this study, the central laboratory will be entrusted with the testing of biomarker samples. About 3.5 mL of venous whole blood will be collected each time.
PK evaluation indicator: JMT103 serum drug concentration | Day 2,15,29 and 3,6,12 months
  Venous blood samples will be collected at the specified time points, about 3.5 mL each time, the actual PK blood collection time should be recorded in the eCRF.
Incidence of JMT103 anti-drug antibodies (ADA) and neutralizing antibodies (NAB) | Day 1,29 and 3,6,12 months
  Blood samples will be collected at the specified time points, about 3.5 ml each time. The JMT103 anti-drug antibody (ADA) in the serum will be tested by electrochemical immunoassay. ADA-positive serum samples will be tested for neutralizing antibodies (NAB).
Types and proportions of adverse events | From signing the informed consent form to 6 months after the last administration
  An adverse event (AE) can be any unfavorable and unanticipated signs (including abnormal laboratory findings), symptoms, or diseases temporally related to the used (study) drug, regardless of whether it is related to the drug or not. A serious adverse event (SAE) refers to any adverse event that meets one of the following criteria:
  Leading to death; Life-threatening; Requiring hospitalization or prolongation of hospitalization; Permanent or severe disability or loss of function; Congenital abnormalities or birth defects; Other significant medical events judged by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Chi Y, Li Y, Cheng Q, Cai H, Zeng Y, Sheng H, Song B, Li H, Shen L, Li M, Xing Y, Cheng M, Ma Y, Wang D, Zhu M, Lu W, Yan S, Zhang X, Yuan J, Yang B, Li J, Wang J, Wu Z, Xia W. Efficacy and safety of narlumosbart, an anti-RANKL monoclonal antibody, in postmenopausal women with osteoporosis: a multi-center, randomized, double-blind, placebo- and active-controlled, phased II study. EClinicalMedicine. 2025 Jul 4;85:103329. doi: 10.1016/j.eclinm.2025.103329. eCollection 2025 Jul. PMID 40686685